CLINICAL TRIAL: NCT00830752
Title: Understanding Alexithymia
Brief Title: Neurobiological, Neuropsychological,Linguistic and Gestural Processes and Phenomena in Individuals With Alexithymia
Acronym: ALEX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Isabella Heuser, Charite
Other Study IDs: ALEX 2009
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Alexithymia
Keywords: alexithymia
MeSH Terms: conditions — Affective Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The syndrome of extremely restricted emotional competence, alexithymia, was originally conceptualized in psychoanalytic research and is now empirically and experimentally studied in clinical psychology and psychological medicine within the context of emotion regulation using neuroscientific techniques. Alexithymia refers to an individual's inability or impaired ability to name or express feelings and to distinguish them from the physical consequences of an acute or chronic stress reaction. Modern "brain-body-interface" research suggests that alexithymia represents a complex deficiency in cognitive processing and emotional regulatory processes. The neurobiological basis is assumed to be a preconscious, automatic and involuntary information transfer to the amygdalae of acquired representations of emotional contents stored in ventromedial prefrontal cortical areas.

Alexithymia is not just "emotional coldness", i.e. a limited emotionality, but essentially the detachment of feelings from language. In alexithymia the link between affective phenomena and language, understood as media-supported sign practices, is insufficient or even absent.

The purpose of our observational study is to better understand the neurobiological and neuropsychological as well as linguistic and gestural processes and determinants of this phenomenon

ELIGIBILITY:
Inclusion Criteria:

* scoring high on the TAS-20

Exclusion Criteria:

* personal history of a mental disorder
* currently mentally ill

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 70 individuals between the ages of 18 and 60 years, both genders, who score high on an alexithymia questionaire (TAS-20) and who are otherwise emotionally and physically healthy. Individuals are sampled via newspaper and poster advertisements throughout the greater metropolitan area of Berlin, Germany
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Charite-Dept. of Psychiatry-Campus Benjamin Franklin, Berlin, Germany